CLINICAL TRIAL: NCT00344500
Title: Management of Antipsychotic Medication Associated Obesity
Brief Title: Healthy Lifestyles for Mentally Ill People Who Have Experienced Weight Gain From Their Antipsychotic Medications
Acronym: MAMAO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D3925-R
Record Dates: First submitted 2006-06-22; First posted 2006-06-26 (Estimated); Results first posted 2015-05-18 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes; Obesity; Weight Gain
Keywords: Antipsychotic; Bipolar; Diabetes; Mental Illness; Nutrition; Obesity; Schizoaffective; Schizophrenia; Weight Gain; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Weight Gain; Mental Disorders; Schizophrenia; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Usual Care
- Lifestyle Balance (Active Comparator): Behavioral Weight Loss Program
  Interventions: Behavioral: Behavioral Weight Loss Program

INTERVENTIONS:
Behavioral: Behavioral Weight Loss Program — Patients randomized to the behavioral weight loss program (Lifestyle Balance Program) will do the following: -Meet with their psychiatrist and a nutritionist who will go over diet recommendations with the patient
  * Be given a 7% weight loss goal
  * Be assisted in obtaining a 500 calorie reduction per day
  * Exercise for at least 30 min/day, at least 5 days a week
  * Maintain weekly food and exercise diaries
  * Be quizzed on their knowledge of healthy eating habits and nutrition
  Other Names: Lifestyle Balance Program
  Arms: Lifestyle Balance

SUMMARY:
This program aims to help Veterans who take antipsychotic medications lose weight. The investigators use a program based on the American Diabetes Association's "Diabetes Prevention Program," and the investigators have modified it to fit the lifestyles of people with mental illness. All participants are educated about nutrition and cutting down fat intake, how and when to exercise, and the causes of diabetes and how to prevent it. Participants must be Veterans who live within one hour of the West Los Angeles VA hospital.

DETAILED DESCRIPTION:
Rationale: The focus of this project is to develop a strategy to combat medication associated weight gain, the most problematic side effect of the newer antipsychotic medications. Improvements in long-term health outcomes might then be expected to change quality of life, promote treatment adherence, rehabilitative potential, and decrease resource utilization.

Procedures:

Half of the patients will randomized to the behavioral weight loss program (Lifestyle Balance Program) and do the following: Meet with their psychiatrist and a nutritionist who will go over diet recommendations with the patient Given a 7% weight loss goal Assisted in obtaining a 500 calorie reduction per day Asked to exercise for at least 30 min/day, at least 5 days a week Maintain weekly food and exercise diaries Be quizzed on their knowledge of healthy eating habits and nutrition

The other half of the patients will be randomized to "Usual Care" and will:

Receive pamphlets about Lifestyle Balance, starting exercise, and general nutritional information regarding food pyramids and the amount of calories in fast foods.

Be encouraged to exercise and eat a healthy diet Not receive classes on nutrition or exercise Be seen on the same schedule as the experimental group, in order to equalize contact time.

After six months, if patients in the "usual care group" wish to participate in the more rigorous behavioral weight loss program they will be given that opportunity.

Visits:

Time Line:

Each subject will be followed for one year. Healthy Lifestyles courses will take eight weeks to complete. Visits will be monthly for the remaining 12 months Enrollment: 120 patients Course of study: October 2005-October 2008

At Beginning and Termination:

Informed Consent (at start of study only) Psychiatric interviews and assessments Physical Examination Framingham risk assessment for cardiovascular disease Electrocardiogram Lipid Profile, fasting glucose, Hemoglobin A1C

At Each Visit:

Vitals, weight, waist circumference, BMI, and % Fat Food and exercise diaries will be reviewed

At Month One and Month Six:

Lipid Profile, fasting glucose, Hemoglobin A1C Electrocardiogram Psychiatric assessments

At Month Nine:

Lipid Profile, fasting glucose, Hemoglobin A1C Electrocardiogram

Clinical Care:

All patients will continue their clinical care with their current psychiatrist and general physician. Medications will not be manipulated for the purpose of this study.

Incentives:

The group participating in the behavioral intervention program will receive rewards for achieving weight loss goals and be given incentives such as a pedometer and Slimfast meal replacements.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran
* Diagnosis of psychotic disorders, schizophrenia, schizoaffective disorder and bipolar illness
* Age 18-70
* Clinically determined to require ongoing treatment with Second Generation Antipsychotics (SGA) such as olanzapine, risperidone, quetiapine, ziprasidone, aripiprazole, clozapine
* Experienced weight gain since treatment with SGA's
* Inpatient or outpatient at the West Los Angeles VA
* Competent to sign informed consent

Exclusion Criteria:

* Have recently been diagnosed with schizophrenia (less than 1 year)
* Are pregnant or breast feeding a baby
* Have a medically unstable condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-10; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Ames, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

REFERENCES:
- [Background] Guzik LH, Wirshing DA. Behavioral weight loss classes for patients with severe mental illness. Psychiatr Serv. 2007 Nov;58(11):1498. doi: 10.1176/ps.2007.58.11.1498. No abstract available. PMID 17978266
- [Result] Erickson ZD, Mena SJ, Pierre JM, Blum LH, Martin E, Hellemann GS, Aragaki DR, Firestone L, Lee C, Lee P, Kunkel CF, Ames D. Behavioral interventions for antipsychotic medication-associated obesity: a randomized, controlled clinical trial. J Clin Psychiatry. 2016 Feb;77(2):e183-9. doi: 10.4088/JCP.14m09552. PMID 26930534
- [Derived] Tully A, Smyth S, Conway Y, Geddes J, Devane D, Kelly JP, Jordan F. Interventions for the management of obesity in people with bipolar disorder. Cochrane Database Syst Rev. 2020 Jul 20;7(7):CD013006. doi: 10.1002/14651858.CD013006.pub2. PMID 32687629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 225 volunteers were screened November 2005 to August 2008 from Veterans Hospital psychiatric clinics in West Los Angeles, USA.
Pre-assignment Details: 122 volunteers met the inclusion criteria, signed the informed consent document, and completed the baseline screening assessments prior to randomization to study groups.
Groups:
- Usual Care: Usual Care control group
- Lifestyle Balance: Weight management education and counseling
  Behavioral Weight Loss Program: Patients randomized to the behavioral weight loss program (Lifestyle Balance Program) will do the following: -Meet with their psychiatrist and a nutritionist who will go over diet recommendations with the patient
  * Be given a 7% weight loss goal
  * Be assisted in obtaining a 500 calorie reduction per day
  * Exercise for at least 30 min/day, at least 5 days a week
  * Maintain weekly food and exercise diaries
  * Be quizzed on their knowledge of healthy eating habits and nutrition
- Changeover: Participants originally randomized to Usual Care who were allowed to change over to Lifestyle Balance at month 6 per their request.
Period: Overall Study
Arm/Group | Usual Care | Lifestyle Balance | Changeover
Started | 48 | 60 | 14
Completed | 25 | 25 | 12
Not Completed | 23 | 35 | 2
Not completed — Adverse Event | 6 | 2 | 0
Not completed — Lost to Follow-up | 5 | 13 | 1
Not completed — Withdrawal by Subject | 7 | 10 | 0
Not completed — Protocol Violation | 4 | 7 | 1
Not completed — Not Noted | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Participants (14) randomized to Usual Care group who later elected to change over to Lifestyle Balance were excluded from statistical analysis.
Groups:
- Lifestyle Balance: Weight management education and counseling
- Total: Total of all reporting groups
Arm/Group | Usual Care | Lifestyle Balance | Total
Number analyzed (Participants) | 48 | 60 | 108
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.58 (9.1) | 49.67 (6.9) | 49.63 (7.9138)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 42 | 54 | 96
Race/Ethnicity, Customized [Number; unit: participants]
  African American or Black | 24 | 25 | 49
  Asian or Pacific Islander | 0 | 2 | 2
  Caucasian, White | 19 | 24 | 43
  Hispanic, Latino, or Spanish Origin | 3 | 6 | 9
  Native American or Alaska Native | 0 | 0 | 0
  Mixed Heritage or Other | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 48 | 60 | 108
Living Situation [Number; unit: participants]
  Own Home | 0 | 1 | 1
  Rental Home/Apt | 6 | 16 | 22
  With Relatives | 2 | 1 | 3
  Board and Care | 40 | 42 | 82
  Homeless | 0 | 0 | 0
Marital Status [Number; unit: participants]
  Married | 8 | 4 | 12
  Single/Cohabiting | 24 | 27 | 51
  Divorced/Widower | 16 | 29 | 45
Education Level [Number; unit: participants]
  No diploma | 3 | 5 | 8
  HS Diploma/GED | 36 | 47 | 83
  Bachelor's or Equivalent Degree | 9 | 6 | 15
  Higher Professional Degree | 0 | 2 | 2
Occupation [Number; unit: participants]
  Paid Work | 3 | 6 | 9
  Unpaid Work | 3 | 1 | 4
  None | 42 | 53 | 95
Medical Comorbidity [Number; unit: participants]
  Hypertension | 27 | 33 | 60
  Dyslipidemia | 23 | 32 | 55
  Diabetes | 11 | 15 | 26
  Metabolic Syndrome | 25 | 40 | 65
  Obesity | 32 | 40 | 72
  Required Exercise Tolerance Test | 5 | 7 | 12
Diagnosis per the Structured Clinical Interview for the Diagnostic and Statistical Manual [Number; unit: participants]
  Schizophrenia | 28 | 21 | 49
  Schizoaffective | 8 | 12 | 20
  Bipolar | 9 | 23 | 32
  Other | 3 | 4 | 7
Antipsychotic (Weight Gain Risk) [Number; unit: participants]
  Olanzapine/Clozapine (High) | 11 | 5 | 16
  Risperidone/Quetiapine (Med) | 20 | 24 | 44
  Aripiprazole/Ziprasidone (Low) | 7 | 21 | 28
  Other | 3 | 2 | 5
  Multiple | 7 | 8 | 15
Length of Psychiatric Illness [Mean (Standard Deviation); unit: years] | 20.5 (11.8) | 18.86 (11.8) | 19.5889 (11.7732)
Age of Onset of Psychiatric Illness [Mean (Standard Deviation); unit: years] | 28.21 (10.12) | 30.47 (11.5) | 29.4656 (10.917)
Baseline Psychopathology Ratings [Mean (Standard Deviation); unit: units on a scale] — Brief Psychiatric Rating Scale: Symptom survey, score range 18 - 126, best to worst.
  Clinical Global Impression: Rates overall psychiatric symptom severity, scored 1-6, best to worst.
  Hamilton Depression Rating Scale: Score range 0 - 78, best to worst.
  Heinrichs Quality of Life Scale: Score range 0-132, worst to best.
  Self-Assessment of Illness Questionnaire: Rates mental health and weight, score range 32 - 128, best to worst.
  Antipsychotics Side-effects Checklist: Score range 17-34, worst to best.
  Motivational Interview to Assess Stage of Change: Scored 0-5, worst to best.
  units on a scale
    Brief Psychiatric Rating Scale, Total | 33.4 (8.0) | 34.9 (8.8) | 34.2333 (8.4483)
    Clinical Global Impression Rating | 3.4 (0.8) | 3.4 (0.8) | 3.4 (0.7963)
    Hamilton Depression Rating Scale, Total | 10.0 (5.9) | 12.7 (7.4) | 11.5 (6.8776)
    Heinrichs Quality of Life Scale, Total | 54.7 (18.9) | 61.1 (22.4) | 58.2556 (21.0662)
    Self-Assessment of Illness Questionnaire, Total | 76.6 (9.18) | 79.1 (9.4) | 77.9889 (9.3433)
    Antipsychotics Side-effects Checklist, Total | 26.2 (3.7) | 25.6 (3.7) | 25.8667 (3.6948)
    Motivational Interview to Assess Stage of Change | 2.9 (0.7) | 2.9 (0.7) | 2.9 (0.6967)
Body Weight [Mean (Standard Deviation); unit: kg] | 106.7 (15.6) | 105.3 (21.0) | 105.9222 (18.7231)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.3 (4.8) | 34.1 (5.3) | 34.1889 (5.0615)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 119.1 (11.4) | 117.1 (14.5) | 117.9889 (13.19)
Percent Body Fat [Mean (Standard Deviation); unit: percentage] | 30.2 (6.6) | 30.8 (5.7) | 30.5333 (6.0941)
Framingham Hard Coronary Heart Disease [Mean (Standard Deviation); unit: Percent] — 10-year risk estimate of developing hard coronary heart disease
  Percent | 10.8 (7.4) | 11.2 (5.8) | 11.0222 (6.5301)
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic | 123.5 (11.9) | 126.7 (13.3) | 125.2778 (12.7394)
  Diastolic | 82.4 (10.6) | 83.1 (10.4) | 82.7889 (10.4459)
Laboratory Tests [Mean (Standard Deviation); unit: mm/dL]
  Glucose | 114.6 (60) | 103.9 (38.6) | 108.6556 (49.3093)
  HDL Cholesterol | 37.5 (9.1) | 37.3 (8.9) | 37.3889 (8.9477)
  Triglycerides | 161.5 (101.4) | 161.3 (117.9) | 161.3889 (110.368)
  LDL Cholesterol | 114.2 (36.1) | 111 (30.9) | 112.4222 (33.1885)
  Total Cholesterol | 184.9 (43.8) | 178.9 (38.1) | 181.5667 (40.6457)
Microalbumin/Creatinine [Mean (Standard Deviation); unit: mgMA/gCrt] | 13.8 (26.7) | 16.12 (39.7) | 15.0889 (34.4026)

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight
Description: Average weight of subjects attending each of the first 8 weekly visits and the 10 monthly visits which followed, per study group.
Time Frame: Weekly/Monthly, up to 1 year
Population: All subjects who enrolled in this research program. Subjects were assessed weekly, when able. Since some were not able to do every weekly assessment, N varies weekly, and the weekly assessments below are the means of the number of subjects out of the total in the group who were assessed at that point.
Measure: Mean (Standard Deviation); unit: Pounds
Groups:
- Usual Care (UC): Usual Care control group
- Lifestyle Balance (LB): Behavioral Weight Loss Program
Arm/Group | Usual Care (UC) | Lifestyle Balance (LB)
Number analyzed (Participants) | 48 | 60
Pounds
  Week 0 (n=47, 60) | 235.22 (34.51) | 232.1 (46.3)
  Week 1 (n=44, 56) | 235.95 (35.33) | 233.41 (46.1)
  Week 2 (n=42, 50) | 232.3 (33.56) | 233.34 (47.78)
  Week 3 (n=38, 45) | 235.98 (35.88) | 233.54 (42.91)
  Week 4 (n=41, 47) | 236.89 (36.03) | 237.84 (51.64)
  Week 5 (n=34, 43) | 235.99 (37.94) | 234.79 (45.95)
  Week 6 (n=38, 41) | 237.88 (37.84) | 237.38 (52.9)
  Week 7 (n=36, 42) | 235.3 (36.54) | 235.5 (52.73)
  Week 8 (n=39, 43) | 236.8 (37.11) | 237.65 (51.67)
  Week 9 (n=0, 1) | NA (NA) — Data collection at this point only occured in one exceptional case. | 251 (0)
  Week 12 (n=39, 36) | 238.2 (36.72) | 237.54 (51.59)
  Week 17 (n=36, 34) | 236.81 (38.09) | 236.9 (52.7)
  Week 21 (n=36, 36) | 238.56 (39.92) | 235.97 (52.46)
  Week 26 (n=31, 34) | 236.26 (41.24) | 234.11 (54.47)
  Week 30 (n=28, 30) | 236.94 (45.59) | 236.23 (58.26)
  Week 34 (n=26, 28) | 239.3 (48.37) | 236.53 (59.64)
  Week 38 (n=26, 28) | 233.23 (43.56) | 230.21 (48.04)
  Week 43 (n=24, 25) | 238.61 (46.43) | 228.25 (48.65)
  Week 48 (n=26, 24) | 238.31 (46) | 229.94 (50.6)
  Week 52 (n=25, 25) | 238.54 (48.09) | 228.39 (51.95)
Statistical Analysis 1: Comparison: Usual Care (UC) vs Lifestyle Balance (LB); General Linear Mixed Model (GLMM) used to illustrate the magnitude of difference between slopes for major outcomes for two hypothetical participants with identical baseline characteristics over 12 months; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Predicted trajectory of mean weight change between matched UC and LB subjects over 12 months (treatment*time interaction: F(1,1275)=68.75, p<.01)

2. Primary Outcome: Change in Predicted Trajectory of Mean BMI Per GLMM Analysis
Description: General Linear Mixed Model (GLMM) is a full information maximum likelihood approach that permits inclusion of all available data and provides unbiased parameter estimates even if there are missing data under the condition that data are missing at random. The GLMM approach assumes that every patient is on a specific trajectory over time and that both the slope and the shape of this trajectory are a potential function of group membership or other person-level covariates. Using a likelihood ratio test, we compared different options to model these trajectories and found a linear model, which assumes that the same rate of change is maintained over the whole study, provided a good fit to the data. We used a linear model of the average rate of change over time (slope) for all comparisons. To illustrate the magnitude of difference between slopes for major outcomes, we report the estimated difference at 12 months between two hypothetical participants with identical baseline characteristics.
Time Frame: 12 months
Measure: Number; unit: kg/m^2
Arm/Group | Usual Care (UC) | Lifestyle Balance (LB)
Number analyzed (Participants) | 48 | 60
kg/m^2 | 0.6 | -1.7

3. Primary Outcome: Change in Predicted Trajectory of Mean Body Fat Percentage Per GLMM Analysis
Description: Computed as % body fat at 12 month - % body fat at baseline. General Linear Mixed Model (GLMM) is a full information maximum likelihood approach that permits inclusion of all available data and provides unbiased parameter estimates even if there are missing data under the condition that data are missing at random. The GLMM approach assumes that every patient is on a specific trajectory over time and that both the slope and the shape of this trajectory are a potential function of group membership or other person-level covariates. Using a likelihood ratio test, we found a linear model, assuming the same rate of change throughout the study, provided a good fit to the data compared to other models. We used a linear model of the average rate of change over time (slope) for all comparisons. To illustrate the magnitude of difference between slopes for major outcomes, we report the estimated difference at 12 months between two hypothetical participants with identical baseline characteristics.
Time Frame: 12 months
Measure: Number; unit: Body Fat Percentage Change
Arm/Group | Usual Care (UC) | Lifestyle Balance (LB)
Number analyzed (Participants) | 48 | 60
Body Fat Percentage Change | 1.5 | -2

ADVERSE EVENTS:
Time Frame: Four (4) years, between November 2005 and October 2009.
Arm/Group | Usual Care | Lifestyle Balance | Changeover
Serious Adverse Events (participants affected / at risk) | 8/48 | 9/60 | 1/14
Other Adverse Events (participants affected / at risk) | 1/48 | 0/60 | 1/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=48) | Lifestyle Balance (N=60) | Changeover (N=14)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0)
Bell's Palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Staph Aureus Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Prescription Medication Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant Pancreatic Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Exacerbated Psychosis (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Pancreatitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Syphilis Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neurotoxic Chemical Exposure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Neurological effect to wood varnish fumes
Exacerbated Mania (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Exacerbated Depresssion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=48) | Lifestyle Balance (N=60) | Changeover (N=14)
Chest/rib pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations to our study were its single-site recruitment yielding subjects mostly male and all veterans, limiting of statistical power by control subjects allowed to join treatment group resulting in exclusion from data, and a high dropout rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes